CLINICAL TRIAL: NCT04092764
Title: Feasibility Study for Electroacupuncture for Chemotherapy- Induced Peripheral Neuropathy (CIPN) Using a Point-Of-Nerve Conduction Device (NeuroMetrix) and the Rydel-Seiffer Tuning Fork
Brief Title: Feasibility Study for Electroacupuncture for Chemotherapy- Induced Peripheral Neuropathy (CIPN)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-20022
Record Dates: First submitted 2019-09-13; First posted 2019-09-17 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy
Keywords: Numbness; Pain; Tingling; Reduced sense of touch; Reduced proprioception; Sensory Neuropathy
MeSH Terms: conditions — Hypesthesia; Pain; Paresthesia | interventions — Electroacupuncture

STUDY DESIGN:
Intervention Model Description: Participants with Sensory Neuropathy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Participants Receiving Electroacupuncture (Experimental): Participants will receive electroacupuncture for 30 minutes once per week for a total of 3 weeks.
  Interventions: Device: Electroacupuncture; Device: NeuroMetrix; Device: Rydel-Seiffer tuning fork

INTERVENTIONS:
Device: Electroacupuncture — Participants will receive electroacupuncture for 30 minutes once per week for a total of 3 weeks. The acupoints will be stimulated by the electroacupuncture machine with alternating frequencies in order to induce endorphins at different points in the nervous system. Frequencies between 2 Hz and 100 Hz will be utilized. Sterile single-use needles will be placed at Ba Feng, four points on the dorsum of each foot between the digits. KI2 (Rang Gu), a point located at the soles of the feet and SP-4 (Gongsun) will also be needled per recommendation of our acupuncturist. A total of 12 needles will be used per participant.
Device: NeuroMetrix — The NeuroMetrix is a point-of-care conduction device that will be used to measure peripheral neuropathy
Device: Rydel-Seiffer tuning fork — The level of periphal neuropathy will be measured by vibration detection using a Rydel-Seiffer graduated tuning fork placed on the dorsum of the right great toe between the nail and the distal interphalangeal joint. The two arms of the 128 Hz tuning fork are fitted with calibrated weights at the ends, and as the amplitude decreases, the intersection of the triangles moves upward on the weight. This test will be performed three times and a mean of the scores calculated. Vibration sensation is lost sooner in CIPN, which means that lower scores are associated with increased CIPN

SUMMARY:
The purpose of the study is to determine the validity of a point-of-care nerve conduction device (NeuroMetrix) and Rydel-Seiffer tuning fork in assessing the level of peripheral neuropathy in patients with chemotherapy-induced peripheral neuropathy (CIPN). Chemotherapy-induced peripheral neuropathy (CIPN) is a common, persistent toxicity among patients who receive chemotherapy. It is characterized by a variety of sensory and motor symptoms such as numbness, tingling, reduced sense of touch, reduced proprioception (awareness of your limb and body position in space), pain, weakness, balance disturbances, and deficits in motor skills.

ELIGIBILITY:
Inclusion Criteria:

* Must have undergone chemotherapy with taxane and/or platinum agent
* Presence of numbness, paresthesias, loss of deep tendon reflexes, or other symptoms in the lower extremities those were absent prior to treatment with neurotoxic chemotherapy.
* Three or more months status post platinum containing chemotherapy completion
* Grade ≥1 Level of CIPN that is determined by the NCI Common Toxicity Criteria for Adverse Events.

Exclusion Criteria:

* Peripheral neuropathy from causes other than chemotherapy, such as documented
* a. Nerve compression (carpal tunnel syndrome, sciatica, etc)
* b. Previously known leptomeningeal carcinomatosis
* c. Evidence of disease in the brain or spine by prior imaging
* Comorbidities with documented pre-existing neuropathy prior to the chemotherapy such as
* a. Diabetes (HbA1c 6.5% or greater)
* b. HIV
* c. Multiple myeloma
* d. Alcoholism
* Pain medication dosing, including opioids, anti-convulsants, and anti- depressantshas been increased due to worsening symptoms less than in the two weeks prior to study registration
* Current use of acupuncture (manual or electro acupuncture)
* Pregnancy
* Cardiac issues (AHA class 3 or greater)
* Pacemaker or an imbedded neural stimulator
* Full therapeutic anticoagulation or a INR > 1.4
* Currently undergoing chemotherapy with a platinum agent or have received a platinum chemotherapy agent in the past 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-01-23 (Actual); Primary Completion 2021-11-09 (Actual); Study Completion 2021-11-11 (Actual)

PRIMARY OUTCOMES:
Accessing Level of Peripheral Neuropathy | Baseline to 30 days after 3 week treatment sessions
  Participants with chemotherapy-induced peripheral neuropathy (CIPN) will have their level of periphal neuropathy assessed with the Rydel-Seiffer Tuning Fork while using a point-of-care conduction device (NeuroMetrix). The level of periphal neuropathy will be measured by vibration detection using a Rydel-Seiffer graduated tuning fork placed on the dorsum of the right great toe between the nail and the distal interphalangeal joint. The two arms of the 128 Hz tuning fork are fitted with calibrated weights at the ends, and as the amplitude decreases, the intersection of the triangles moves upward on the weight. This test will be performed three times and a mean of the scores calculated. Vibration sensation is lost sooner in CIPN, which means that lower scores are associated with increased CIPN.

SECONDARY OUTCOMES:
Quality of life Improvement measured with FACT/GOG-NTX Questionnaire | Baseline to 30 days after 3 week treatment sessions
  Quality of life improvement with electroacupuncture treatment will be measured using the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity questionnaire (FACT/GOG-NTX). The FACT/GOG-NTX questionnaire uses 37 questions with a scale ranging from 0-4, with 0 being Not at All and 4 being Very Much.
Quality of life Improvement measured the Neuropathic pain scale (NPS) | Baseline to 30 days after 3 week treatment sessions
  The NPS has 3 questions using a scale ranging from 0-100 with 0 being No Numbess Sensation to 100 being Worst Numbness Imaginable. The NPS also has 10 Yes or No questions about pain. A score of 1 is given to each question answered Yes and a score of 0 to each questions answered No. The total score is calculated as the sum of the 10 questions, and the cut off value for the diagnosis of neuropathic pain is 4/10.

CONTACTS AND LOCATIONS:
Overall Officials: Hye Sook Chon, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2019-08-23): https://cdn.clinicaltrials.gov/large-docs/64/NCT04092764/ICF_000.pdf